CLINICAL TRIAL: NCT07026890
Title: The Value of Virtual Reality in the Care of Elderly People With Psychomotor Disadaptation Syndrome: a Randomised Controlled Trial of Mixed Efficacy and Implementation vs. Conventional Rehabilitative Care
Brief Title: The Benefits of Virtual Reality in the Care of Elderly People With Psychomotor Disadaptation Syndrome
Acronym: VIR-AGE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: DIPANDA 2024
Record Dates: First submitted 2025-06-10; First posted 2025-06-18 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Psychomotor Disadaptation Syndrome

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: conventional rehabilitation + 3 virtual reality sessions (Experimental)
  Interventions: Other: Evaluation visits; Other: Rehabilitation sessions; Other: Virtual reality sessions
- Control: conventional rehabilitation + 3 additional rehabilitation sessions (Active Comparator)
  Interventions: Other: Evaluation visits; Other: Rehabilitation sessions; Other: Additional rehabilitation sessions

INTERVENTIONS:
Other: Evaluation visits — 3 assessment visits (initial (V1), intermediate (V2) and final (V3).
  A series of motor assessments carried out by the physiotherapist:
  * Timed Up and Go Test (TUG)
  * 10 m walk test (TM10)
  * Functional Reach Test (FRT)
  * Minimum Motor Test (TMM)
  * 10 m walk test combined with a verbal task such as naming different animals
Other: Rehabilitation sessions — Usual treatment: 4 to 5 rehabilitation sessions per week, each lasting 45 minutes.
Other: Virtual reality sessions — 3 virtual reality sessions per week, each lasting 30 minutes.
  Arms: Experimental: conventional rehabilitation + 3 virtual reality sessions
Other: Additional rehabilitation sessions — 3 additional rehabilitation sessions per week. These sessions correspond to standard rehabilitation sessions.
  Arms: Control: conventional rehabilitation + 3 additional rehabilitation sessions

SUMMARY:
Psychomotor Disadaptation Syndrome (PMDS) is characterised by a deterioration in postural function, gait and psychomotor automatisms in the elderly. It is often associated with falls and can manifest itself as retropulsion, gait abnormalities, neurological disorders and psycho-behavioural problems. For the majority of these patients, a stay in a geriatric medical and rehabilitation centre is necessary, enabling an objective assessment of these disorders and multi-professional care, including physiotherapists, occupational therapists and adapted physical activity teachers, aimed at restoring safe movement and motor independence. However, rehabilitation relies on traditional exercises that are limited, repetitive and sometimes far removed from everyday activities. Technological innovations such as virtual reality (VR) offer opportunities to improve care by creating immersive environments that reproduce real-life situations. VR could thus help to rehabilitate the motor problems associated with MS.

The aim of the VIR-AGE project is to study the clinical benefits of VR in the rehabilitation of hospitalised elderly people suffering from PMDS in terms of functional deficits, particularly motor deficits.

The study will take place at the Centre gériatrique Champmaillot of the CHU Dijon Bourgogne. A total of 50 patients with SPDM will take part.

The total duration of your participation is 5 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Person who has given written consent
* Person aged ≥ 65 years;
* With a proven diagnosis of motor maladjustment syndrome;
* Hospitalised in a geriatric care unit;
* Able to understand a simple instruction and answer a closed question;

Exclusion Criteria:

* Person not affiliated to or not benefiting from a social security scheme
* Person subject to a legal protection measure (curatorship, guardianship)
* Person subject to a judicial protection measure
* An adult who is incapable or unable to give consent
* Persons with epilepsy, kinetosis or known claustrophobia Persons unable to understand simple instructions for carrying out tests
* Anyone with a severe visual and/or hearing impairment
* Any person with a behavioural disorder (agitation, aggressiveness)
* Any person with a severe walking or balance problem that makes motor exercises unsuitable
* Anyone with a pathology, injury, wound or severe deformity to the head or cervical spine
* Any person suffering from severe vertigo, diagnosed at the discretion of the investigating doctor
* Inability to use arm for pointing
* Persons susceptible to migraines
* Non-French speakers
* Anyone with an inter-pupillary distance outside the range of possible helmet adjustments

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-07-16 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Change in 'Timed Up and Go' time between initial and final assessment | 5 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Dijon Bourgogne, Dijon, France